CLINICAL TRIAL: NCT02075892
Title: Acute Effects of a Mushroom Blend on Oxygen Kinetics, Aerobic Power and Time to Fatigue
Brief Title: Mushroom Blend on Oxygen Kinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Scivation, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 14-0062
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-08

CONDITIONS: Oxygen Utilization; Oxygen Kinetics
Keywords: cordyceps, aerobic capacity, exercise performance, fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mushroom Blend (Active Comparator): 4 grams daily; oral; 7 and 21 days
  Interventions: Dietary Supplement: Mushroom Blend
- Placebo (Placebo Comparator): 4 grams maltodextrin, oral, 7 and 21 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mushroom Blend — Scivation
  Other Names: Cordyceps
  Arms: Mushroom Blend
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Purpose: To determine the acute effects of a mushroom blend vs. placebo on oxygen kinetics, aerobic power and time to fatigue in healthy adults.

DETAILED DESCRIPTION:
Participants: Twenty-eight, healthy, active, recreationally-trained adults ages 18-35.

Procedures (methods): All subjects will report to the Applied Physiology Laboratory in Fetzer Rm 025 for phase I of the study for a total of 7 visits. A randomly selected subset of 8 participants will continue to phase II, and return to the lab for an additional 3 visits to evaluate feasibility. Visit 1 will consist of a physical, enrollment and consenting. Visits, 2, 3, and 4 will be separated by a minimum of 24 hours. During visit 2, participants will perform a maximal oxygen consumption (VO2max) test on a cycle ergometer. During visit 3 participants will be asked to complete a 6-minute oxygen kinetics test on a cycle ergometer; lactate threshold and oxygen saturation will be measured at baseline, minutes 2, 3 and 6 during the 6 min ride. During visit 4, participants will perform a 3-minute critical power (CP) test and will provide a saliva sample, to be measured for cortisol levels, immediately prior to and after the CP test. Following visit 4, participants will be randomly assigned, in a double-blind fashion, to either a placebo or mushroom blend treatment group. Participants in the placebo and treatment groups will be asked to consume 2 servings, 3 times daily for 7 days. Following supplementation, participants will return to the laboratory for visits 5-7, each of which will be separated by a minimum of 24 hours. The same protocol performed during visits 2-4 will be repeated in the same order for visits 5-7; the VO 2max test, the 6 min oxygen kinetics test, and the CP test with a pre and post saliva sample. The randomly selected subset of 8 participants will continue into phase II (n=4 for treatment; n=4 for placebo). During phase II, the 8 participants in the placebo and treatment groups will be asked to consume 2 servings, 3 times daily for 14 additional days to determine feasibility of a longer supplementation phase. Following supplementation, the same protocol performed during visits 2-4 will be repeated in the same order for visits 8-10, each of which will be separated by a minimum of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Participant has been involved in exercise program for a minimum of one year prior to recruitment (≥ 3 d/wk)
* Participant is able to exercise (i.e. no existing musculoskeletal injury)
* Participant is willing and able to comply with the protocol
* Participant is apparently healthy and free from disease, as determined by a health history questionnaire and physical
* Participant agrees to abstain from smoking, caffeine, tobacco, and alcohol before testing days
* Participant agrees to abstain from exercise 24 hours prior to each testing visit
* Participant is not allergic to mushrooms

Exclusion Criteria:

* Participant has a BMI ≤ 28 kg/m² (pre-screening inclusion)
* Having a history of medical or surgical events that may significantly affect the study outcome, including cardiovascular disease, metabolic, renal, hepatic, or musculoskeletal disorders
* Participant is using, or has used one of the following dietary supplements within 12 weeks prior to enrollment: Beta-alanine, Creatine, Carnosine or Taurine
* Participant has lost or gained greater than ten pounds within the previous 3 month
* Participant is currently enrolled in another clinical trial.
* Participant has a known allergy or sensitivity to any ingredient in the test product or placebo (determined from health history questionnaire)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Oxygen kinetics | during a 6 min
  oxygen uptake and utilization using indirect calorimetry during a 6 min steady-state exercise bout
Critical Power | during a 3 min
  3 min all-out cycling test to measure anaerobic and aerobic performance

SECONDARY OUTCOMES:
Lactate | baseline, 2min, 3min, 6min (pre-post supplementation)
Cortisol | during a 6 min
Maximal Oxygen Consumption | during a graded exercise test to exhaustion
  oxygen consumption and utilization using indirect calorimetry during a graded exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina
Locations (1):
- Applied Physiology Laboratory, Fetzer Hall, Chapel Hill, North Carolina, United States